CLINICAL TRIAL: NCT06197672
Title: Chimeric Antigen Receptor T Cell Redirected to Target CD4 Positive Relapsed Refractory AML as a Bridge to Allogeneic Stem Cell Transplant
Brief Title: Chimeric Antigen Receptor T Cell Redirected to Target CD4 Positive Relapsed Refractory Acute Myeloid Leukemia (AML ) as a Bridge to Allogeneic Stem Cell Transplant
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Huda Salman (Other)
Collaborators: iCell Gene Therapeutics (Industry)
Responsible Party: Sponsor-Investigator, Huda Salman, Director, Hematologic Malignancies Service and Director, CAR T Cellular Therapy Program, Indiana University
Organization: Indiana University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CTO-IUSCCC-0851
Record Dates: First submitted 2023-12-14; First posted 2024-01-09 (Actual); Last update posted 2026-01-22 (Actual); Status verified 2026-01

CONDITIONS: Acute Myeloid Leukemia
Keywords: Acute Myeloid Leukemia; T Cell; Cell Therapy; CAR T; Chimeric Antigen Receptor Therapy
MeSH Terms: conditions — Leukemia, Myeloid, Acute

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (Experimental): Redirected autologous T cells transduced with the anti-CD4 lentiviral vector (referred to as "CD4CAR" cells)
  Interventions: Biological: CD4CAR

INTERVENTIONS:
Biological: CD4CAR — CD4CAR cells transduced with a lentiviral vector to express the single-chain variable fragment (scFv) nucleotide sequence of the anti-CD4 molecule derived from humanized monoclonal ibalizumab and the intracellular domains of CD28 and 4-1BB co-activators fused to the CD3ζ T-cell activation signaling domain administered by IV infusions as a single dose

SUMMARY:
This study is designed as a single arm open label traditional Phase I, 3+3, study of CD4-redirected chimeric antigen receptor engineered T-cells (CD4CAR) in patients with relapsed or refractory AML. The study will evaluate safety in this patient population and also the presence of efficacy signal described by elimination of residual disease to qualify patients for stem cell transplant.

DETAILED DESCRIPTION:
The study will be performed as a dose-escalation protocol. The investigators expect to recruit 20 subjects at Indiana University with an expected dropout rate of 25% primarily due to rapid progression or death and screen and or manufacturing failure. Taking this into account, the investigators expect to treat 15 patients. The study will utilize autologous CD4CAR T-cells that are engineered to express a chimeric antigen receptor (CAR) targeting CD4 that is linked to the cluster of differentiation 28 (CD28), 4-1BB, cluster of differentiation 3-zeta (CD3ζ) signaling chains (third generation CAR). about 70% of AML with monocytic differentiation and 37% of all the rest express CD4 on their blasts.

At entry, disease status will be staged. Qualifying subjects will be leukapheresed to obtain large numbers of peripheral blood mononuclear cells (PBMC) for the manufacturing. Next, participants will receive conditioning chemotherapy. If tumor burden is sufficiently reduced (screening step), participants will receive CD4CAR cells by infusion on Day 0 of treatment.

If the disease progresses during the manufacturing period participants may be excluded from the study or an attempt to bridge for disease control will be offered. Minimal chemotherapy to keep the disease under control in the meanwhile is allowed if deemed necessary by investigators.

A single dose of CD4CAR transduced T cells will consist of the cell number for the dose level to be infused.

Post-infusion monitoring of CD4CAR T-cells: Subjects will have blood drawn for cytokine levels, CD4CAR Transgene Copy Number (PCR) and flow cytometry in order to evaluate the presence of CD4CAR cells on days 0, 1, 3, 5, 7, 14, and 28 following infusion (or as clinically needed). Cytokines levels will be evaluated per schedule above in addition to and as needed every 8 +/- 2 hours as feasible if/when Cytokine Release Syndrome, CRS, occurs and until resolution. Active monitoring of fungal and viral infections during treatment while utilizing standard prophylaxis recommended for HIV-positive patients with T-cell aplasia and those undergoing allogeneic stem cell transplant. Investigators plan to collect data about clinicoradiologic measurements of residual tumor burden starting on day 7 and weekly afterward until Day 28 and then monthly for 6 months. This will be followed by quarterly clinical evaluations for the next two (2) years with a medical history, physical examination, and comprehensive blood testing. After these short- and intermediate-term evaluations are performed, these patients will enter a rollover study to assess for disease-free survival (DFS), relapse, and the development of other health problems or malignancies where follow-up will be up to twice a year by phone and a questionnaire for an additional thirteen (13) years. The treating physician will decide to proceed with allogeneic or autologous transplant when needed.

Dose of CD4CAR description: the main objective of this study is to establish a recommended dose and/or schedule of CD4CAR. The guiding principle for dose escalation in phase I is to avoid unnecessary exposure of patients to sub-therapeutic doses (i.e., to treat as many patients as possible within the therapeutic dose range) while preserving safety and maintaining rapid accrual. Investigators will use the rule-based traditional Phase I "3+3" design for the evaluation of safety. Based on lab experience in mice the starting dose (dose level 1) for the first cohort of three patients in phase I portion of the study will be 8x10^5 cells. The dose escalation or de-escalation will follow a modified Fibonacci sequence as below.

If more than one patient out of the first cohort of three patients in dose level 1 experience dose limiting toxicity (DLT), the trial will be placed on hold. If zero or one out of three patients in the first cohort of dose level 1 experience DLT, three more patients will be enrolled at dose level 1; the dose escalation continues until at least two patients among a cohort of six patients experience DLT (i.e., ≥33% of patients with a DLT at this dose level)

If one of the first three patients in dose level 1 experiences a DLT, three more patients will be treated at dose level 1.

If none of the three patients or only one of the 6 patients in the dose level 1 experiences a DLT, the dose escalation continues to the dose level 2 If one of the first three patients in dose level 2 experience a DLT, three more patients will be treated at dose level 2 If none of the three patients or only one of the 6 patients in the dose level2 experiences a DLT, the dose escalation continues to the dose level 3 If one of the first three patients in dose level 3 experiences a DLT, three more patients will be treated at dose level 3 If none of the three patients or only one of the 6 patients in the dose level 3 experiences a DLT, dose level 3 will be declared the maximum tolerated dose (MTD) and will be used as the recommended phase II dose (RP2D) for the phase II portion of the study.

In summary, the dose escalation continues until at least two patients among a cohort of six patients experience DLT (i.e., ≥33% of patients with a DLT at that dose level). The recommended dose for phase II trials is defined as one dose level below this toxic dose level. Since some grade 3 and possibly 4 toxicities are highly likely to be reversible, grade 3 infectious, hematological and vascular toxicities will not be considered DLTs mandating dose reduction. Also allergic or infusion-related reactions ≤ grade 3 will not be counted as DLTs. There will be no intra-patient dose escalation or reduction.

To allow for full spectrum toxicity duration evaluation and reporting, no patients within the same or a different cohort will be initiated on lymphodepleting chemotherapy sooner than 28 days from the initiation date of the preceding patient.

ELIGIBILITY:
Inclusion Criteria:

1. ≥ 12 years old at the time of informed consent
2. Ability to provide written informed consent and HIPAA authorization.
3. Diagnosis of AML that is CD4+ and must have failed standard induction/ first line treatment such as intensive induction or less intensive hypomethylation and venetoclax first line. In the specific case of azacitidine and venetoclax (aza/ven), BM biopsy for response assessment on days 21-28 of first cycle. If disease progression by increasing number of blasts is documented, patient will be eligible. If no morphologic remission (persistent BM blasts above 5%) but evidence of efficacy exists, a second cycle without interruption will be given with the goal of achieving morphologic remission and repeat BM biopsy on days 21-28 of this cycle. If residual disease or disease progression is captured, then they will be considered refractory and will qualify for this trial. This is unless the patient now qualifies for a more intensive induction therapy that they did not qualify for when aza/ven was initially chosen as first-line treatment. Given the low response rate for aza/ven in the RR-AML, CR of only 13%, this combination would not be a prerequisite to qualify for the study.
4. If these patients who fail first line treatment have an FDA approved treatment options available (including targeted and non-targeted treatment) for a second line treatment, they do not qualify for the trial until they also are deemed nonresponsive to those. If an approved second line is not available, patients will be eligible after first line failure.
5. Creatinine clearance of > 60ml/min (or otherwise non clinically significant, per study investigator)
6. alanine aminotransferase/ aspartate aminotransferase ALT/AST < 3 x ULN
7. Bilirubin < 2 x ULN (UPPER LIMIT OF NORMAL)
8. Pulmonary Function Test (PFT) with a DIFFUSE LUNG CAPACITY , DLCO, of ≥ 60% (if not completed within 6 months from Day 0)
9. Adequate echocardiogram with EJECTION FRACTION, EF, of ≥50%
10. Adequate venous access for apheresis and no other contraindications for leukapheresis
11. Confirmation of a bone marrow donor for post CD4CAR transplant to proceed to transplant if eligible post treatment.

Exclusion Criteria:

1. CD4 negative AML
2. Pregnant or lactating women. The safety of this therapy on unborn children is not known. Female study participants of reproductive potential (see definition below) must have a negative serum or urine pregnancy test prior to initiation of conditioning chemotherapy, per research sites' clinical policy.
3. Uncontrolled active infection necessitating systemic therapy.
4. Active hepatitis B hb, or hepatitis C, HC, infection. Active hepatitis C is defined as the hepatitis C antibody is positive while quantitative HCV RNA results exceed the lower detection limit.

   Note the following subjects will be eligible:
   * Subjects with a history of hepatitis B but have received antiviral therapy and have non-detectable viral DNA for 6 months prior to enrollment are eligible.
   * Subjects seropositive for HBS antibodies due to hepatitis B virus vaccine with no signs or active infection (Negative HBs Ag, HBc and HBe Ags) are eligible.
   * Subjects who had hepatitis C but have received antiviral therapy and show no detectable hepatitis C virus (HCV) viral RNA for 6 months are eligible.
   * If hepatitis C antibody test is positive, then patients must be tested for the presence of antigen by reverse transcription-polymerase chain reaction (RT-PCR) and be hepatitis C virus ribonucleic acid (HCV RNA) negative.
5. Concurrent use of systemic glucocorticoids in greater than replacement doses or steroid dependency defined in rheumatological and pulmonary diseases as uninterrupted corticosteroid intake for more than a year at a dosage of 0.3 mg/kg/day or greater, and where the underlying disease worsens on temporary stoppage of steroid therapy, with symptoms of steroids withdrawal (eg, lethargy, headache, weakness, pseudo rheumatism, emotional disturbances, etc) precipitated by the temporary stoppage unless tapering can occur safely without compromising the underlying disease, the withdrawal tolerance and can happen in a timeframe appropriate to enroll in this trial without safety concerns

   Subjects who receive daily corticosteroids in replacement doses can be included in the study. The replacement doses are defined as following:
   1. Hydrocortisone 25mg/day or less
   2. Prednisone 10mg/day or less
   3. Dexamethasone 4mg or less Note: Recent or current use of inhaled glucocorticoids is not exclusionary, as this route pertains extremely minimal systemic penetration
6. Any previous treatment with any gene therapy products
7. Any uncontrolled active medical disorder that would preclude participation as outlined in the opinion of the treating investigator and/or Principal Investigator
8. HIV infection
9. Subjects who have received or will receive live vaccines within 30 days before the first experimental cell treatment. Inactivated seasonal flu vaccination is allowed.
10. Subjects with active autoimmune diseases who need systematic treatments (such as disease modifying agents, corticosteroids, and immunosuppressive drugs) during the last year.

    Note: Replacement therapy (thyroxine, insulin, or physiological corticosteroid replacement therapy (up to10 mg of oral daily prednisone or equivalent in hydrocortisone and dexamethasone) to treat adrenal dysfunction or pituitary dysfunction) is not considered as systematic therapy. Subjects who need inhalation corticosteroid therapy can be included in this trial. Subjects with vitiligo or in long-term remission of pediatric asthma or allergic diseases can be included in this trial.
11. Subjects with a history of mental disorders or drug abuse that may influence treatment compliance.
12. Active malignancy not related to AML that has required therapy in the last 3 years or is not in complete remission. Exceptions to this criterion include successfully treated non-metastatic basal cell or squamous cell skin carcinoma, or prostate cancer that does not require therapy. Other similar malignant conditions may be discussed with and permitted by the Principal Investigator.
13. Participation in another clinical study with an investigational product within the past 6 months provided patient was in fact given that experimental treatment, just being enrolled and treated is not a disqualifier.

Eligibility for Conditioning Chemotherapy:

1. Specific organ function criteria for cardiac, renal, and liver function must be similar to initial inclusion values.
2. Review of co-morbidities to confirm no major changes in health status (examples of major changes include heart attack, stroke, and any major trauma).
3. Planned infusion does was successfully manufactured and met release criteria.
4. Negative pregnancy testing (if applicable).

Eligibility for CD4CAR infusion:

1. Afebrile and not receiving antipyretics, and no evidence of active infection. If fever is attributed to underlying disease, it will not disqualify.
2. Specific organ function criteria for cardiac, renal, and liver function must be similar to initial inclusion values. The following tests do not need repeated: an echocardiogram if within 6 weeks of initial assessment, and the PFT if completed within 6 months from Day 0.
3. If previous history of corticosteroid chemotherapy, subject must be off all but adrenal replacement doses 3 days before the CD4CAR infusion.

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-03-19 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2042-12-31 (Estimated)

PRIMARY OUTCOMES:
1. Dose finding: Maximum tolerated dose (MTD) is defined as one dose level lower than the Dose Limiting Toxicity (DLT) of the CD4CAR in AML. Optimal dose is highest safe dose that produces the most response. | Day 0 through Day 28 post-infusion
  In this traditional phase 1 dose escalation, cohorts of three subjects will be treated on a dose level that will be incremented to next dose level if no dose limiting toxicities (DLT) were reported or expanded if a DLT is documented.
Persistence and biologic behavior of CD4CAR as measured by a. Serial blood and marrow sampling to detect CD4CAR over time post infusion. b. Serial testing for CD4CAR proliferation, differentiation and polarization if feasible overtime after infusion. | Day 0 Through Day28 post infusion
  The persistence of the CAR through day 28 and possibly longer if detected by D28. This will be performed by flow to assess for the CD3+/Fab2+ cell population The phenotype of the CAR will be determined by flow as well, to look for Tcm phenotype
3. Determine the influence of CD4CAR on T regs | Day 0 through Day 28
  1. Examine the efficacy of CD4CAR on changing the frequency of T regs subpopulation after CD4CAR infusion as compared to their frequency prior to treatment.
  2. Determine the impact of the change in T regs and MDSCs abundance on objective response to CD4CAR.
Determine the influence of CD4CAR on myeloiod derived suppressor cells, MDSCs | Day 0 through Day 28
  Examine the efficacy of CD4CAR on changing the frequency of MDSCs subpopulation

SECONDARY OUTCOMES:
Determine mLSCs frequency before and after the CD4CAR infusion | Baseline through Day 30
  Participants' blood will be tested by flow cytometry to determine the ability of CD4CAR to target Monocytic Leukemia Stem Cells (mLSCs).
Quantification of CD4CAR associated cytokines | Baseline through Day 30
  Participants blood will be examined for cytokine level changes according to time points as described in the protocol.
Describe disease response using European LeukemiaNet (ELN) 2022 recommendation | Baseline through Day 30
  Treatment is intended to reduce the disease burden enough to qualify patients for stem cell transplant through either elimination of residual disease or minimizing that to being acceptable to transplant consideration. For response evaluation of the frequency of successful bridging to transplant, European LeukemiaNet (ELN) 2022 recommendation will be applied.

CONTACTS AND LOCATIONS:
Overall Officials: Huda Salman, MD, PhD, Principal Investigator — Indiana University
Locations (4):
- United States (4):
  - University of Miami Sylvester Comprehensive Cancer Center, Miami, Florida
  - Indiana University Melvin and Bren Simon Comprehensive Cancer Center, Indianapolis, Indiana
  - Riley Hospital for Children, Indianapolis, Indiana
  - The University of Texas MD Anderson Cancer Center, Houston, Texas